CLINICAL TRIAL: NCT05715021
Title: Randomized Trial Evaluating First Time Shoulder Dislocation: Surgery vs Conservative Care
Brief Title: RCT Evaluating First Time Shoulder Dislocation
Acronym: REDUCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Moin Khan, Associate Professor and Orthopaedic Surgeon, McMaster University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REDUCE
Record Dates: First submitted 2023-01-18; First posted 2023-02-06 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Shoulder Dislocation; Sport Injury; Anterior Dislocation
MeSH Terms: conditions — Shoulder Dislocation

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial with Embedded Non-randomized Cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Bankart repair + Remplissage (randomized cohort) (Experimental): Arthroscopic repair of anterior capsulo-labral structures
  Interventions: Procedure: Bankart + Remplissage Procedure
- Conservative treatment (randomized cohort) (No Intervention): Non surgical intervention
- Bankart repair + Remplissage (non-randomized cohort) (Experimental): Arthroscopic repair of anterior capsulo-labral structures
  Interventions: Procedure: Bankart + Remplissage Procedure
- Conservative treatment (non-randomized cohort) (No Intervention): Non surgical intervention

INTERVENTIONS:
Procedure: Bankart + Remplissage Procedure — Participants will undergo arthroscopic stabilization.
  Arms: Bankart repair + Remplissage (non-randomized cohort); Bankart repair + Remplissage (randomized cohort)

SUMMARY:
The primary objective of the pilot study is to assess the feasibility of a definitive trial to determine the effect of arthroscopic soft tissue stabilization vs. non-operative management on the risk of recurrent anterior dislocation rates and functional outcomes following in patients presenting with a first-time dislocation (FTD) over a 24-month period.

DETAILED DESCRIPTION:
Background

The shoulder is the most commonly dislocated joint in the body with a global incidence that ranges from 15 to 25 per 100 000 people. It is estimated that approximately 70 000 shoulder dislocations occur annually in the United States. In North America, a sampling of individuals presenting with shoulder dislocations to US emergency departments identified an overall incidence rate in the United States of 24 (95% confidence interval, 20.8 to 27.0) per 100,000 person-years and a maximum incidence rate (47.8 [95% confidence interval, 41.0 to 54.5]) occurring in those between the ages of twenty and twenty-nine years. A review of shoulder reductions performed in emergency rooms in Ontario, Canada between 2002 and 2010 identified 719 dislocations affecting primarily young patients with a median age of 35 years and 74% male. The incidence density rate of shoulder dislocations was found to be 23/100,000 person-years and highest among young males (98/100,000 person-years).

Recurrence mainly occurs in the first 2 years after the first anterior shoulder dislocation event, and recurrent instability significantly affects quality of life, sport, and professional activities.4 Epidemiologic data suggests that younger patients are at significantly higher the risk of recurrence. In a prospective study of 252 patients by Robinson et al, the recurrence rate after 5 years reached 86.6% in patients aged 15 to 20 years, 73.8% in patients between 21 and 25 years of age, and 46.8% in patients between 26 and 30 years of age. Participation in contact and overhead throwing sports and higher sporting levels also increases the risk of recurrence.

Management options in patients with a first-time shoulder dislocation include non-operative and operative approaches.

Anterior dislocations often injure the anterior and inferior glenoid labrum, described as the Bankart lesion. This lesion was observed arthroscopically in 94% to 100% of patients and often result in long-term instability. Thus, there is debate as to whether arthroscopic Bankart repair should be routinely performed in patients after a first-time anterior shoulder dislocation.

Historically, non-operative treatment has been the most common method of managing first-time dislocations. Additionally, for young athletes, non-operative treatment is often advocated in season to allow for rapid return to sport despite concerns regarding recurrent instability. Owens et al. demonstrated that non-operative management of an in-season shoulder dislocation can allow a return to sports in as little as 7 to 21 days, however early return increased the risk for further instability episodes, particularly in throwing or overhead athletes. Another study found that although 88.6% of 15- to 25- year-old athletes undergoing non-operative management returned to sport, 71.4% experienced recurrent dislocations. Given recent research and limited available evidence over the past 10 years, surgical management has been suggested as a potentially more reliable method to prevent further dislocations and improve patient outcomes when compared with non-operative management.

Arthroscopic soft tissue repair (Bankart repair) has become increasingly popular given the advancement in surgical technique allowing for a minimally invasive and reliable improvement in instability with a low risk of complication. The high recurrence rate in younger patients may justify offering surgical treatment after the first episode of FTD. A recent systematic review by Hurley et al. found arthroscopic Bankart repair resulted in a 7-fold lower recurrence rate and a higher rate of return to play than conservative management.

Current surgical practice however is generally consideration for surgical management only if further instability or recurrence has occurred. Recurrence however increases a patient's risk of further injury to the humeral head and glenoid - potentially resulting in poorer outcomes. Although some studies show arthroscopic treatment after first episodes of FTD in younger patients results in low dislocation rates, such treatment is not universally recognized or practiced. Additionally, concern regarding overtreatment exists - a network meta-analysis by Kavaja et al. found for patients 47% of patients receiving non-surgical management did not experience further shoulder dislocations. Significant controversy therefore exists regarding optimal management of this widespread condition.

Need for a Pilot Study Prior to a Large Trial A pilot study is needed prior to a large trial to determine the feasibility of a larger trial in terms of ability to recruit across clinical sites, adherence to study protocol and ability to follow participants for 24 months.

Primary objective is to examine the feasibility of a larger trial. Feasibility objectives include:

1. Ability to recruit across multiple clinical sites.
2. Ability to follow participants for 24 months.
3. Ability to operate on patients within 3 months following enrollment.
4. Assessment of crossovers.

Secondary objectives: compare arthroscopic capsuloligamentous repair vs. non-surgical intervention on:

1. Recurrent shoulder dislocations up to 24 months' post-treatment.
2. Symptoms of instability without dislocation up to 24 months post treatment.
3. Clinical outcomes measured by Western Ontario Shoulder Instability (WOSI) Index, American Shoulder and Elbow Society (ASES) score, Shoulder Activity Scale, EQ-5D, Visual Analog Scale (VAS) Pain Score, and Patient Satisfaction questionnaire.
4. Physical examination: range of motion, stability.
5. Return to previous level of activity and work.
6. Safety, shoulder-related complications and serious adverse events.

The investigators propose a multi-centre pilot RCT to compare the effect of arthroscopic surgical stabilization (Bankart procedure) and non-operative management (physical therapy) in patients with a post-traumatic first-time shoulder anterior dislocation. Eligible and consenting participants will be followed-up by the site for 24 months. Outcomes will be assessed at 6 weeks, 6 months, 12 months, and 24 months post-treatment. Since the decision between surgery and conservative management may be heavily influenced by patient preference, we will also embed a prospective non-randomized cohort within this RCT to capture all patients who would be eligible for the study but refuse to be randomized. These patients will choose to either undergo arthroscopic stabilization or non-operative management to treat their FTD and will be followed the same way as the randomized cohort. This study design not only ensures maximal participation but is also more generalizable to the real world where preferences might play a role in shared decision-making.

For participants who agree to be randomized, eligible and consenting participants will be randomized to one of two treatment groups:

* Arthroscopic capsuloligamentous repair (Bankart +/- Remplissage Procedure; intervention group)
* Non-operative management (physical therapy; control group)

Participants who agree to participate in the non-randomized arm of the study will not be randomized. Their treatment preference will be noted at baseline.

Once participants have provided informed consent, baseline demographics, relevant medical history, and details regarding their diagnosis will be collected from the participant, the attending surgeon, their medical record and through physical examination. Participants will also complete The Western Ontario Shoulder Instability Index (WOSI), the American Shoulder and Elbow Surgeons questionnaire (ASES), EQ-5D, patient satisfaction scale at the time of enrolment.

After surgery, surgical and peri-operative details will be collected from the attending surgeon and the participant's medical records. Adverse events occurring during the surgical procedure or perioperative period will also be documented.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ages 14-40 years;
2. Diagnosis of first-time shoulder anterior dislocation having occurred within the past 3 months confirmed either by radiographic evidence or documented reduction of anterior shoulder dislocation as well as physical examination eliciting unwanted glenohumeral translation with reproduction of symptoms;
3. Provision of informed consent.

Exclusion Criteria:

1. Patients that cannot undergo surgery or anesthesia;
2. Patients with concomitant injuries (rotator cuff tear, fracture)
3. Previous shoulder surgery;
4. Patients that will likely have problems with maintaining follow-up or are incarcerated;
5. Epilepsy/seizure disorder;
6. Pregnancy;
7. Diagnosis of multidirectional instability;
8. Bony glenoid defect (bony Bankart) >10% as measured on preop imaging;
9. Dislocation without trauma, in a context of hyper laxity or atraumatic instability;
10. Cases involving litigation or workplace insurance claims (e.g., WSIB).

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07-12 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment Feasibility | 10 months
  Number of patients recruited
Follow-up | 2 years
  Proportion of participants followed at two years
Surgery within 3 months of enrollment | 3 months
  Ability to operate on patients within 3 months following enrollment
Crossovers | 2 years
  Assessment of crossovers between groups

SECONDARY OUTCOMES:
Rate of Recurrence Dislocation | 2 years
  Rate of recurrent dislocation between patients randomized to arthroscopic surgical repair and those receiving conservative treatment.
Rate of Instability | 2 years
  Rate of symptomatic instability/positive apprehension sign between patients randomized to arthroscopic surgical repair and those receiving conservative treatment.
Clinical Outcome - shoulder function | 2 years
  Measured by Western Ontario Shoulder Instability (WOSI) Index. The final score ranges from 0 (best possible score - the patient is experiencing no decrease in shoulder related quality of life) to 2100 (worst score - signifies extreme distress in shoulder related quality of life).
Clinical Outcome | 2 years
  Measured by American Shoulder and Elbow Society (ASES) score. Scores range from 0 to 100 with a score of 0 indicating a worse shoulder condition and 100 indicating a better shoulder condition.
Clinical Outcome - Quality of Life | 2 years
  Measured by EQ-5D (EuroQol-5 Dimension). The EQ-5D comprises five questions on mobility, self care, pain, usual activities, and psychological status with three possible answers for each item (1=no problem, 2=moderate problem, 3=severe problem. A summary index with a maximum score of 1 can be derived from these five dimensions by conversion with a table of scores. The maximum score of 1 indicates the best health state, by contrast with the scores of individual questions, where higher scores indicate more severe or frequent problems.
Clinical Outcome - shoulder activity | 2 years
  Measured by Shoulder Activity Scale.The activity rating is a numerical sum of scores for five activities rated on a five-point frequency scale from never performed (0 points) to daily (4 points).
Clinical Outcome - pain | 2 years
  Measured by Visual Analog Scale (VAS) Pain Score. 0 - no pain, 10 - the worst pain
Clinical Outcome - patient satisfaction | 2 years
  Measured by Patient Satisfaction questionnaire. 0 - least satisfied, 10 - most satisfied
Range of motion | 2 years
  Assessed in forward flexion, abduction, external rotation and internal rotation.
Rate of participants with risk of having recurrent shoulder instability | 2 years
  Measured by apprehension-relocation physical examination maneuver (positive or negative)
Rate of participants that return to previous level of activity | 2 years
  Return to previous level of activity and sport (self reported)
Return to work | 2 years
  Duration of work stoppage if applicable
Adverse events | 2 years
  Rate of major and minor shoulder-related complications and serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Moin Khan, MD, Principal Investigator — McMaster University
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No